CLINICAL TRIAL: NCT04803474
Title: Turner And Klinefelter Treatment Target Study. Improving Endocrine Treatment by Linking Biochemical Parameters to Morbidity and Quality of Life in Patients With Turner and Klinefelter Syndrome
Brief Title: Turner And Klinefelter Treatment Target Study
Acronym: TAKTT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: dr. Laura C. G. de Graaff-Herder (Other)
Responsible Party: Sponsor-Investigator, dr. Laura C. G. de Graaff-Herder, Principal investigator, Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Other Study IDs: NL65814.078.18
Record Dates: First submitted 2020-07-02; First posted 2021-03-17 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Klinefelter Syndrome; Turner Syndrome
MeSH Terms: conditions — Klinefelter Syndrome; Turner Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Klinefelter: Patients with Klinefelter syndrome
  Interventions: Diagnostic Test: Measurement of blood values, questionnaire scores and measurements of hormone levels in hair
- Turner: Patient with Turner syndrome
  Interventions: Diagnostic Test: Measurement of blood values, questionnaire scores and measurements of hormone levels in hair

INTERVENTIONS:
Diagnostic Test: Measurement of blood values, questionnaire scores and measurements of hormone levels in hair — Measurement of blood values, questionnaire scores and measurements of hormone levels in hair

SUMMARY:
Rationale: Health related Quality of life (HRQoL) is impaired in patients with Turner and Klinefelter syndrome (TS and KS). It is unknown what the optimal endocrine treatment target values are that maximize HRQoL in patients with these syndromes. Therefore the relation between HRQoL and biochemical parameters will be studied in large cohorts of patients with TS and KS. This information will give essential insight that will help to improve endocrine treatment and HRQoL in these patients.

Research objectives: To explore the relationship between biochemical parameters and HRQoL in patients with TS and KS.

Hypothesis: Biochemical parameters are related to HRQoL in patients with TS and KS.

Study design: Cross-sectional, observational, multicentre study Study population: Patients with KS or TS, 18 years or older Methods and procedures: To measure fatigue the Checklist Individual Strength (CIS-20) will be used, for QoL the 5-level EQ-5D (EQ-5D-L5) will be used and for stress the Perceived Stress Scale (PSS) and hair cortisol levels. For patients with KS the anxiety scale from the Liebowitz social anxiety scale (LSAS) will be used to measure social anxiety. To measure the long-term exposure to testosterone in KS patients, testosterone concentrations in hair will be measured. For patients with KS, all questions from the questionnaires will be discussed orally during a visit to the outpatients clinic. One extra tube of blood and a strand of hair will be collected during routine blood withdrawal. All other variables are already part of the standard patient care and are available in patient records. For patients with TS all information including the questionnaires and laboratory values is already available and will be collected from clinical records.

Main study parameters/endpoints: The relationship between different hormonal parameters and HRQoL as measured by questionnaires. The main hormonal parameter that will be investigated in KS is testosterone in hair. For patients with Turner syndrome, free thyroxine (FT4), thyroid stimulating hormone (TSH) and liver enzymes, which have already been collected, will be investigated. The relationships between the EQ-5D-L5 score and testosterone in hair (in patients with KS) and thyroid hormone status (in patients with TS) are the primary outcomes.

DETAILED DESCRIPTION:
Rationale: Health related Quality of life (HRQoL) is impaired in patients with Turner and Klinefelter syndrome (TS and KS). It is unknown what the optimal endocrine treatment target values are that maximize HRQoL in patients with these syndromes. Therefore the relation between HRQoL and biochemical parameters will be studied in large cohorts of patients with TS and KS. This information will give essential insight that will help to improve endocrine treatment and HRQoL in these patients.

Research objectives: To explore the relationship between biochemical parameters and HRQoL in patients with TS and KS.

Hypothesis: Biochemical parameters are related to HRQoL in patients with TS and KS.

Study design: Cross-sectional, observational, multicentre study

Study population: Patients with KS or TS, 18 years or older Methods and procedures: To measure fatigue the Checklist Individual Strength (CIS-20) will be used, for QoL the 5-level EQ-5D (EQ-5D-L5) will be used and for stress the Perceived Stress Scale (PSS) and hair cortisol levels. For patients with KS the anxiety scale from the Liebowitz social anxiety scale (LSAS) will be used to measure social anxiety. To measure the long-term exposure to testosterone in KS patients, testosterone concentrations in hair will be measured. For patients with KS, all questions from the questionnaires will be discussed orally during a visit to the outpatients clinic. One extra tube of blood and a strand of hair will be collected during routine blood withdrawal. All other variables are already part of the standard patient care and are available in patient records. For patients with TS all information including the questionnaires and laboratory values is already available and will be collected from clinical records.

Main study parameters/endpoints: The relationship between different hormonal parameters and HRQoL as measured by questionnaires. The main hormonal parameter that will be investigated in KS is testosterone in hair. For patients with Turner syndrome, free thyroxine (FT4), thyroid stimulating hormone (TSH) and liver enzymes, which have already been collected, will be investigated. The relationships between the EQ-5D-L5 score and testosterone in hair (in patients with KS) and thyroid hormone status (in patients with TS) are the primary outcomes.

Objectives:

Primary Objective:

To explore the relationship between thyroid hormone status* and QoL as measured by the EQ-5D-5L in patients with TS.

To explore the relationship between testosterone concentrations in hair and QoL as measured by the EQ-5D-5L in patients with KS.

Secondary Objective(s):

For TS:

The relationship between thyroid hormone status* and the CIS-20 and PSS scores. The relationship between liver enzymes** and the EQ-5D-5L, CIS-20 and PSS scores.

The relationship between hair cortisol levels and the EQ-5D-5L, CIS-20 and PSS scores.

For KS:

The relationship between testosterone concentrations in hair and the CIS-20, LSAS and PSS scores.

The relationship between hair cortisol levels and the EQ-5D-5L, CIS-20, LSAS and PSS scores.

*Variable that consists of the following 6 categories:

* Overt hyperthyroidism (FT4>25pmol/L and TSH<0,4mU/L)
* Overt hypothyroidism (FT4 <11 pmol/L and TSH >4,3 mU/L)
* Subclinical hypothyroidism with TSH <10mU/L (FT4 11-25 pmol/L and TSH 4,3-10mU/L)
* Subclinical hypothyroidism with TSH >10mU/L (FT4 11-25 pmol/L and TSH > 10mU/L)
* Subclinical hyperthyroidism (FT4 11-25 pmol/L and TSH <0,4 mU/L)
* Euthyroidism (FT4 11-25 pmol/L and TSH 0,4- 4,3 mU/L)

  * aspartate aminotransferase (ASAT), alanine aminotransferase (ALAT), alkaline phosphatase (ALP), gamma-glutamyl transpeptidase (GGT), bilirubin, lactate dehydrogenase (LDH)

Study design:

2. STUDY DESIGN This is study is a multicentre cross-sectional cohort study with the Erasmus Medical Centre (EMC), the VU University Medical Centre (VUmc) and the Amsterdam Medical Centre (AMC) as contributing centres. The duration of the study is 26 months.

The following data will be collected: laboratory values, fatigue scores, HRQoL scores, stress-scores, date of birth, age at diagnosis, height, weight, use of medication, genetic background, comorbidities. All information is already available in clinical records for patients with TS. For patients with KS information on HRQoL, fatigue and stress scores needs to be collected. A strand of hair to measure long-term testosterone and cortisol levels in hair and an extra tube of blood for storage will also be collected. This tube of blood could later be used to determine CAGn polymorphism in the androgen receptor, see paragraph below. Patients with KS visit an endocrinologist at the outpatients clinic of the AMC, VUmc or the EMC every one or two years and will be asked all questions of the questionnaires right after their appointment with the endocrinologist. The executive researcher will be present at the outpatients clinic to obtain informed consent and ask all questions. All laboratory values needed are routinely assessed at every visit for standard patient care and will be collected from clinical records afterwards.

2.1 Laboratory values

Laboratory outcomes:

For KS: luteinizing hormone (LH), follicle-stimulating hormone (FSH), testosterone in blood and testosterone and cortisol levels in hair.

For TS: thyroid stimulating hormone (TSH), free T4 (fT4) and liver enzymes: aspartate aminotransferase (ASAT), alanine aminotransferase (ALAT), alkaline phosphatase (ALP), gamma-glutamyl transpeptidase (GGT), bilirubin, lactate dehydrogenase (LDH) and cortisol levels in hair.

2.2 Genotype The classic form of KS, which is present in the 80-90 % of the cases, is defined by a 47,XXY karyotype. Higher-grade aneuploidies (e.g. 48,XXXY or 48,XXYY), structurally abnormal X chromosome (e.g. 47,iXq,Y) or mosaicisms (e.g. 47,XXY/46,XY) make up the remaining 10-20 % of cases.

The most common genetic background in TS patients is a 45,X karyotype, which is present in approximately 60% of TS patients. Around 20% of cases of TS are caused by a mosaicism 45X/46,XX and structural abnormalities chromosome X explain the last 20%. (26) As genetic background influences phenotype, information on karyotype from clinical records will be collected.

2.3 Questionnaires Checklist Individual Strength (CIS-20) To measure fatigue the Checklist Individual Strength (CIS-20) will be used. The CIS-20 consists of 20 questions that measure the amount of fatigue experienced by the subject during the last two weeks. The subject has to indicate on a 7 point Likertscale to what extent each statement applies to him or her. The CIS-20 consists of 4 subscales: subjective fatigue (8 questions), concentration (5 questions), motivation (4 questions) and activity (3 questions). The CIS-20 questionnaire has been validated in several populations and has proven to be a valid and reliable questionnaire for the assessment of fatigue. Utilization of the CIS-20 questionnaire is free, as long a reference to two articles is included in the publication.

5-level EQ-5D (EQ-5D-L5) To assess HRQoL the EQ-5D-L5 questionnaire will be used. This questionnaire consists of two components: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). In the descriptive system the patient is asked to rate how many problems he or she experiences in the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The scores for these five dimensions can be combined to get a number that describes the health state of the respondent. The EQ VAS is also a measure of health outcome. The patient is asked to indicate on a visual analogue scale how good he or she thinks his or her health is. References values for the Dutch general population are available.

Perceived Stress Scale (PSS) To measure stress the PSS questionnaire will be used. The PSS consists of 10 questions that measure the degree of stress experienced by a subject after or during certain events during the preceding month. The PSS has proven to be a valid measure for perceived stress with good psychometric properties.

Liebowitz social anxiety scale (LSAS) To measure social anxiety in patients with Klinefelter syndrome, the LSAS will be used. The LSAS is widely used to measure social anxiety. It consists of two subscales: the scale for anxiety and for avoidance. Respondents are asked to rate their level of fear and avoidance in 24 social situations. Research shows good psychometric properties. Only the scale for anxiety will be used to minimize the burden for the patient.

2.4 Androgen receptor CAGn polymorphism A study by Zitzmann et al. showed an association between androgen receptor CAG repeats and androgen action. KS men with a shorter CAGn length seem to have less gynecomastia, bigger testis and higher bone density. When KS men with a shorter CAGn length receive testosterone replacement therapy, they show a better suppression of LH levels, prostate growth and higher haemoglobin concentrations. However, a more recent study by Valente et al. showed no relevant clinical differences in KS patients due to CAGn length variation on the androgen receptor. Therefore it is currently unclear whether CAG repeats are of clinical importance. Blood samples (buffy coat) will be collected and stored to be able to measure androgen receptor CAG repeats when the role of these CAGn polymorphisms has been clarified.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

For patients with KS: There are no risks associated with participation. All measurements will take place right after a planned visit at the outpatients clinic. All subjects with KS need to answer questions from four questionnaires, which will take about 30 minutes (including collection of informed consent). The biochemical parameters measured are already routinely assessed during the visits to the outpatients clinic. Only one extra tube of blood will be collected and stored. Blood will be collected during blood withdrawal for the assessment of laboratory values needed for standard care. One strand of hair will also be collected.The burden is therefore minimal.

For patients with TS: For patients with TS all information is already available. Therefore there will not be any burden or risk.

There is no direct benefit for the participants, but all patients with KS and TS could benefit from better hormonal treatment in the future due to the results of this study. When the questionnaires indicate severe psychological problems, psychological care will be offered.

ELIGIBILITY:
Inclusion Criteria:

* Klinefelter or Turner syndrome as confirmed by genetic testing
* Sufficient knowledge of the Dutch language to complete the questionnaires
* At least 18 years old

Exclusion Criteria:

* KS: Patients not under treatment in the EMC, AMC or VUmc or no planned visits during the study period
* TS: No laboratory values or no questionnaires available in patient records
* Severe psychiatric or neurologic disorders or other reasons for inability to complete the questionnaires as assessed by the treating physician.
* Failure to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with KS and TS of 18 years or older that visit the outpatients clinic of the EMC, AMC or the VUmc will be included. Approximately 120 KS and 250 TS patients are intended to be included.
Sampling Method: Non-Probability Sample
Enrollment: 370 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
The relationship between thyroid hormone status* and QoL as measured by the EQ-5D-5L in patients with TS. | At study entry (cross-sectional study). There is just one visit per patient. The total study has an approximately duration of 3-4 years.
  thyroid hormone status is a variable that consists of the following 6 categories:
  * Overt hyperthyroidism (FT4>25pmol/L and TSH<0,4mU/L)
  * Overt hypothyroidism (FT4 <11 pmol/L and TSH >4,3 mU/L)
  * Subclinical hypothyroidism with TSH <10mU/L (FT4 11-25 pmol/L and TSH 4,3-10mU/L)
  * Subclinical hypothyroidism with TSH >10mU/L (FT4 11-25 pmol/L and TSH > 10mU/L)
  * Subclinical hyperthyroidism (FT4 11-25 pmol/L and TSH <0,4 mU/L)
  * Euthyroidism (FT4 11-25 pmol/L and TSH 0,4- 4,3 mU/L)
  The range of the EQ-5D-5L is from 0 to 100. A higher score means a better outcome.
The relationship between testosterone concentrations in hair and QoL as measured by the EQ-5D-5L in patients with KS. | At study entry (cross-sectional study). There is just one visit per patient. The total study has an approximately duration of 3-4 years.
  The range of the EQ-5D-5L is from 0 to 100. A higher score means a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Laura de Graaff, MD, PhD, Principal Investigator — Department of Internal Medicine - Endocrinology, Erasmus MC, Rotterdam, the Netherlands
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
Data available upon reasonable request